CLINICAL TRIAL: NCT05624047
Title: The Effect of Breastfeeding Education Via Hybrid Simulation Method in the Antenatal Period on Postpartum Breastfeeding: A Randomized Controlled Trial
Brief Title: The Effect of Breastfeeding Education Via Hybrid Simulation Method in the Antenatal Period on Postpartum Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Sultan OZKAN SAT, Assistant Professor, Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SOZKANSAT
Record Dates: First submitted 2022-11-13; First posted 2022-11-21 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Breastfeeding education using the hybrid simulation method
  Interventions: Behavioral: Breastfeeding education using hybrid simulation method; Behavioral: Routine verbal breastfeeding education
- Control Group (Other): Routine verbal breastfeeding education
  Interventions: Behavioral: Routine verbal breastfeeding education

INTERVENTIONS:
Behavioral: Breastfeeding education using hybrid simulation method — In addition to the verbal breastfeeding training given to the pregnant women assigned to the experimental group, breastfeeding training will be given using the hybrid simulation method consisting of a wearable breast model and standard patient practice.
  Arms: Experimental Group
Behavioral: Routine verbal breastfeeding education — Women in this group will receive oral breastfeeding training, which is routinely given in the pregnant education class and consists of one session.

SUMMARY:
This study aimed to determine the effect of breastfeeding education given to pregnant women by a hybrid simulation method in the antenatal period on postpartum breastfeeding. This study will be carried out in a family health center in Turkey. Breastfeeding education will be given to pregnant women using a hybrid simulation method consisting of a wearable breast model and the standard patient in the intervention group. Women in the control group will receive only routine breastfeeding education.

DETAILED DESCRIPTION:
The research will be conducted as a randomized controlled trial. The stratified block randomization methods will be used to assign women to the intervention and control groups. The personal information form and Breastfeeding Self-Efficacy Scale Short Form (Antenatal) will be implemented to all women before the intervention. Breastfeeding education will be given to pregnant women using a hybrid simulation method consisting of a wearable breast model and the standard patient to support women in breastfeeding and to ensure the continuity of breastfeeding in the postpartum period. Breastfeeding education will be given to women in the 32-36 weeks of pregnancy in the antenatal period. The control group will be received the routine antenatal breastfeeding education given to all women by healthcare personnel as part of the family health center procedures. The Breastfeeding Self-Efficacy Scale Short Form (Postnatal) and the LATCH Breastfeeding Assessment Tool will be administered to women in both the experimental and control groups within the postpartum fifth days and at sixth week postpartum.

ELIGIBILITY:
Inclusion Criteria:

* being between 32-36 weeks of pregnancy
* being primipara or multipara
* being at least literate
* being planning to breastfeed
* agreeing to participate in the study

Exclusion Criteria:

* having a physical or mental health problem that would prevent breastfeeding
* preterm labor (before 37 weeks)
* either mother or baby having a health problem after birth
* being with multiple pregnancy
* being with high-risk pregnancy

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-12 (Actual); Study Completion 2023-08-12 (Actual)

PRIMARY OUTCOMES:
The Breastfeeding Self-Efficacy Scale-Short Form (Antenatal) | Baseline: Between 32 and 36 weeks of pregnancy
  The scale consists of 14 questions and is a five-point Likert type. The lowest score of 14 points and the highest of 70 points are obtained from the scale. The higher the score indicates a higher self-efficacy perception.
The Breastfeeding Self-Efficacy Scale-Short Form (Postnatal) | Postpartum on the fifth day
  The scale consists of 14 questions and is a five-point Likert type. The lowest score of 14 points and the highest of 70 points are obtained from the scale. The higher the score indicates a higher self-efficacy perception.
The Breastfeeding Self-Efficacy Scale-Short Form (Postnatal) | Postpartum 6th week
  The scale consists of 14 questions and is a five-point Likert type. The lowest score of 14 points and the highest of 70 points are obtained from the scale. The higher the score indicates a higher self-efficacy perception.
LATCH Breastfeeding Assesment Tool | Postpartum on the fifth day
  The LATCH Breastfeeding Assesment Tool was developed to objectively evaluate breastfeeding success. LATCH consists of five evaluation criteria. Each criterion is evaluated between 0-2 points. The lowest score that can be obtained from the entire scale is 0 and the highest score is 10. The higher score indicates a higher breastfeeding. success.
LATCH Breastfeeding Assesment Tool | Postpartum 6th week
  The LATCH Breastfeeding Assesment Tool was developed to objectively evaluate breastfeeding success. LATCH consists of five evaluation criteria. Each criterion is evaluated between 0-2 points. The lowest score that can be obtained from the entire scale is 0 and the highest score is 10. The higher score indicates a higher breastfeeding. success.

CONTACTS AND LOCATIONS:
Overall Officials: Sultan Özkan Şat, Dr, Principal Investigator — Bitlis Eren University
Locations (1):
- Bitlis Hüsrevpaşa Family Center, Bitlis, Turkey (Türkiye)